CLINICAL TRIAL: NCT00262236
Title: A Twelve-week, Randomized, Double-blind, Parallel-group, Multicenter, Dose Escalation Study to Evaluate the Efficacy and Safety of Aliskiren Administered Alone and in Combination With Atenolol in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Aliskiren and Atenolol in Adults (>18) With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2304
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Hypertension, Aliskiren, Atenolol, Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
This is a study for people diagnosed with hypertension to compare the safety and effectiveness of aliskiren alone and in combination with atenolol. Each patient will be in the study for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients 18 years of age and older.
2. Patients with essential hypertension.

Exclusion Criteria:

Severe hypertension, Current diagnosis of heart failure, History or evidence of a secondary form of hypertension, Participation in any investigational drug study within one month of planned participation,

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 12 weeks
Diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 12 weeks
Blood pressure of < 140/90 mmHg after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Dietz R, Dechend R, Yu CM, Bheda M, Ford J, Prescott MF, Keefe DL. Effects of the direct renin inhibitor aliskiren and atenolol alone or in combination in patients with hypertension. J Renin Angiotensin Aldosterone Syst. 2008 Sep;9(3):163-75. doi: 10.1177/1470320308096411. PMID 18957387